CLINICAL TRIAL: NCT00113269
Title: Phase 4, Randomized, Open-label, Comparative, Multicenter Study to Assess the Safety and Efficacy of Induction Agents, Alemtuzumab, Basiliximab or Rabbit Anti-thymocyte Globulin in Combination With Tacrolimus, MMF, and a Rapid Steroid Withdrawal in Renal Transplant Recipients
Brief Title: Safety/Efficacy of Induction Agents With Tacrolimus, MMF, and Rapid Steroid Withdrawal in Renal Transplant Recipients
Acronym: INTAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Clinical Trial Registries, Astellas Pharma Global Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-04-003
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Kidney Transplantation
Keywords: Treatment Effectiveness; Treatment Efficacy; Anti-rejection therapy; Immunosuppression; Therapy, antirejection; Renal Transplantation; Transplantation, Kidney; Transplantation, Renal; Grafting, Kidney
MeSH Terms: interventions — Basiliximab; Antilymphocyte Serum; thymoglobulin; Tacrolimus; Alemtuzumab; Mycophenolic Acid; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Alemtuzumab High-Risk Patients (Experimental): Alemtuzumab, tacrolimus, mycophenolate mofetil and steroids; High risk patients: Panel reactive antibody ≥ 20% or re-transplant or African American
  Interventions: Drug: tacrolimus; Drug: alemtuzumab; Drug: mycophenolate mofetil; Drug: steroids
- Conventional High-Risk Patients (Active Comparator): Rabbit anti-thymocyte globulin, tacrolimus, mycophenolate mofetil and steroids; High risk patients: Panel reactive antibody ≥ 20% or re-transplant or African American
  Interventions: Drug: rabbit anti-thymocyte globulin; Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: steroids
- Alemtuzumab Low- Risk Patients (Experimental): Alemtuzumab, tacrolimus, mycophenolate mofetil and steroids; Low risk patients: Panel reactive antibody < 20% and first transplant and non-African American
  Interventions: Drug: tacrolimus; Drug: alemtuzumab; Drug: mycophenolate mofetil; Drug: steroids
- Conventional Low-Risk Patients (Active Comparator): Basiliximab, tacrolimus, mycophenolate mofetil and steroids; Low risk patients: Panel reactive antibody < 20% and first transplant and non-African American
  Interventions: Drug: basiliximab; Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: steroids

INTERVENTIONS:
Drug: basiliximab — IV
  Other Names: simulect
  Arms: Conventional Low-Risk Patients
Drug: rabbit anti-thymocyte globulin — IV
  Other Names: Thymoglobulin
  Arms: Conventional High-Risk Patients
Drug: tacrolimus — oral
  Other Names: Prograf, FK506
Drug: alemtuzumab — Intravenous (IV)
  Other Names: campath
  Arms: Alemtuzumab High-Risk Patients; Alemtuzumab Low- Risk Patients
Drug: mycophenolate mofetil — oral
  Other Names: MMF; CellCept
Drug: steroids — IV and/or oral

SUMMARY:
The purpose of this study is to compare the safety and efficacy of different induction agents (alemtuzumab, basiliximab or rabbit anti-thymocyte globulin) in renal transplant recipients treated with tacrolimus, mycophenolate mofetil (MMF) and a rapid steroid withdrawal.

DETAILED DESCRIPTION:
A 2 arm (1 Active, 1 Active Control) study is to compare the safety and efficacy of different induction agents (alemtuzumab, basiliximab or rabbit anti-thymocyte globulin) in renal transplant recipients treated with tacrolimus, MMF and a rapid steroid withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary or re-transplanted deceased donor kidney or a primary or re-transplanted non-human leukocyte antigen (HLA) living donor kidney (ie., HLA identical or 0 antigen mismatch deceased donor kidneys are allowed).

Exclusion Criteria:

* Patient has previously received an organ transplant other than a kidney
* Patient receiving chronic steroid therapy at time of transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (25):
- United States (25):
  - Birmingham, Alabama
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Livingston, New Jersey
  - New Brunswick, New Jersey
  - Hawthorne, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Danville, Pennsylvania
  - Harrisburg, Pennsylvania
  - Charleston, South Carolina
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Background] Hanaway MJ, Woodle ES, Mulgaonkar S, Peddi VR, Kaufman DB, First MR, Croy R, Holman J; INTAC Study Group. Alemtuzumab induction in renal transplantation. N Engl J Med. 2011 May 19;364(20):1909-19. doi: 10.1056/NEJMoa1009546. PMID 21591943
- See also: Link to Prescribing Information — http://www.astellas.us/docs/prograf.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Started | 76 | 70 | 175 | 180
Received Treatment | 70 | 69 | 164 | 171
Completed | 51 | 48 | 134 | 140
Not Completed | 25 | 22 | 41 | 40
Not completed — Not transplanted, donor issues | 4 | 0 | 2 | 2
Not completed — Not transplanted, recipient issues | 2 | 1 | 7 | 4
Not completed — Early graft loss, technical | 0 | 0 | 2 | 0
Not completed — Death in operating room | 0 | 0 | 0 | 1
Not completed — Did not meet eligibility - pre-treatment | 0 | 0 | 0 | 2
Not completed — Adverse Event | 2 | 7 | 11 | 7
Not completed — Withdrawal by Subject | 4 | 3 | 4 | 2
Not completed — Graft loss | 6 | 6 | 4 | 9
Not completed — Protocol Violation | 1 | 0 | 4 | 2
Not completed — Lost to Follow-up | 2 | 3 | 6 | 3
Not completed — Sponsor elected to discontinue patient | 1 | 0 | 0 | 1
Not completed — Discontinued due to rejection | 0 | 0 | 1 | 0
Not completed — Moved | 0 | 1 | 0 | 3
Not completed — Received pancreas transplant | 0 | 0 | 0 | 2
Not completed — Withdrew consent, Prednisone initiated | 0 | 0 | 0 | 1
Not completed — Did not meet eligibility criteria | 1 | 0 | 0 | 1
Not completed — Unable to return for follow up | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients | Total
Number analyzed (Participants) | 70 | 69 | 164 | 171 | 474
Age, Customized [Number; unit: Participants] — One patient turned 18 years of age during the study.
  Participants
    <18 years | 0 | 0 | 1 | 0 | 1
    Between 18 and 64 years | 66 | 64 | 145 | 146 | 421
    >=65 years | 4 | 5 | 18 | 25 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 49 | 58 | 170
  Male | 37 | 39 | 115 | 113 | 304
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 18 | 20 | 155 | 161 | 354
  Black | 50 | 47 | 2 | 1 | 100
  Asian | 2 | 2 | 5 | 7 | 16
  Other | 0 | 0 | 2 | 2 | 4
Previous Transplant [Number; unit: Participants]
  Yes | 14 | 10 | 2 | 3 | 29
  No | 56 | 59 | 162 | 168 | 445
Type of Transplant [Number; unit: Participants]
  Living related | 21 | 15 | 64 | 74 | 174
  Living non-related | 7 | 11 | 45 | 48 | 111
  Deceased | 42 | 43 | 55 | 49 | 189
Panel Reactive Antibody (PRA) Group [Number; unit: Participants] — PRA is defined as the highest level at time of transplant or 6 months prior to transplant.
  Participants
    Missing | 0 | 1 | 1 | 1 | 3
    0% | 33 | 32 | 134 | 130 | 329
    > 0% - 20% | 14 | 16 | 24 | 39 | 93
    > 20% - 50% | 11 | 7 | 2 | 1 | 21
    > 50% | 12 | 13 | 3 | 0 | 28

OUTCOME MEASURES:

1. Primary Outcome: Patient Incidence of Biopsy-confirmed Acute Rejection (BCAR) at 6 Months
Description: A BCAR is a suspected new rejection w/in 6 mos. of skin closure, confirmed by Banff Grade ≥1A assigned by a pathologist. The Banff 97 classification system is used for interpreting histology of allograft biopsies, including Mild (1A/1B), Moderate (2A/2B) & Severe (3).
  Kaplan Meier analysis was used to estimate % of pts. w/event. Patients w/no event at time of scheduled visit or whose 1st event was after premature discontinuation of study drug/tacrolimus were censored on the scheduled day of a) assessment, b) of premature treatment discontinuation or c) last evaluation, whichever came 1st.
Time Frame: 6 months
Population: The number of participants analyzed per arm represents Full Analysis Set (FAS), which included all patients who were transplanted in the study and received at least 1 dose of tacrolimus and at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 6.2 [0.3 to 12.0] | 9.4 [2.2 to 16.7] | 1.9 [0.0 to 4.0] | 17.5 [11.7 to 23.3]
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.4889, Normal approximation; Analysis based on normal approximation using Greenwood's formula for standard error; differences in event rates = -3.3, 95.305% CI 2-sided [-12.7 to 6.1] — 95.305% Confidence Interval is reported, as adjusted for interim analysis based on normal approximation using Greenwood's formula for standard error
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p < 0.0001, normal approximation; Analysis based on normal approximation using Greenwood's formula for standard error; differences in event rates = -15.7, 95.305% CI 2-sided [-21.9 to -9.4] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Overall Patient Incidence of BCAR
Description: Overall patient incidence of BCAR is defined as a suspected new rejection at any time following skin closure confirmed by a Banff Grade ≥ 1A as assigned by a local pathologist. Incidence is reported as the percentage of patients with BCAR. The Banff 97 scale is a classification system for interpreting histology of allograft biopsies. The grades range from Mild (1A & 1B) to Moderate (2A & 2B) to Severe (3).
  End of Study was defined as the last day of evaluation and could have included bivariate assessments after 36 months.
Time Frame: End of Study (36 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 15.7 | 13.0 | 9.8 | 21.6
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.6533, normal approximation; differences in event rates = 2.7, 95% CI 2-sided [-9.0 to 14.3]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p = 0.0024, normal approximation; differences in event rates = -11.9, 95% CI 2-sided [-19.5 to -4.2]

3. Secondary Outcome: Efficacy Failure
Description: Efficacy Failure is a composite measure of biopsy confirmed acute rejection, graft loss and death. Data is reported as the percentage of patients with Efficacy Failure.
  End of Study was defined as the last day of evaluation and could have included bivariate assessments after 36 months.
Time Frame: End of Study (36 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 22.9 | 29.0 | 15.9 | 24.6
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.4087, normal approximation; differences in event rates = -6.1, 95% CI 2-sided [-20.7 to 8.4]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p = 0.0456, normal approximation; differences in event rates = -8.7, 95% CI 2-sided [-17.2 to -0.2]

4. Secondary Outcome: Clinically Treated Acute Rejection
Description: Clinically treated acute rejection is defined as patient incidence of any rejection (suspected or otherwise) for which treatment was provided. Data is reported as the percentage of patients with Clinically Treated Acute Rejection.
  End of Study was defined as the last day of evaluation and could have included bivariate assessments after 36 months.
Time Frame: End of Study (36 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 22.9 | 21.7 | 12.8 | 26.9
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.8742, normal approximation; differences in event rates = 1.1, 95% CI 2-sided [-12.7 to 15.0]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p = 0.0010, normal approximation; differences in event rates = -14.1, 95% CI 2-sided [-22.5 to -5.7]

5. Secondary Outcome: Time to First BCAR
Description: Time to first BCAR is defined as the number of days from skin closure to the first episode of BCAR.
  End of Study was defined as the last day of evaluation and could have included bivariate assessments after 36 months.
Time Frame: End of Study (36 months)
Population: The number of participants analyzed per arm represents Full Analysis Set (FAS), which included all patients who were transplanted in the study and received at least 1 dose of tacrolimus and at least 1 dose of study drug.
  Only patients who experienced BCAR were included in the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 11 | 9 | 15 | 36
Days | 226 [25 to 1023] | 49 [10 to 769] | 469 [53 to 1065] | 13 [2 to 848]

6. Secondary Outcome: Graft Survival at 12 Months
Description: Graft survival is defined as no graft loss (re-transplant, return to dialysis for more than 30 days or death) with 12 months of skin closure.
  Kaplan Meier analysis was used to estimate percentage of patients with event. Patients with no event by the time of the scheduled visit or whose first event was after premature discontinuation of randomized study drug or tacrolimus were censored on the scheduled day of assessment, on the day of premature treatment discontinuation or last evaluation day, whichever came first.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 95.6 | 92.1 | 97.5 | 95.1
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.4134, normal approximation; Analysis based on normal approximation using Greenwood's formula for standard error; differences in event rates = 3.5, 95% CI 2-sided [-4.8 to 11.7]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p = 0.2459, normal approximation; Analysis based on normal approximation using Greenwood's formula for standard error; differences in event rates = 2.4, 95% CI 2-sided [-1.7 to 6.5]

7. Secondary Outcome: Overall Graft Survival
Description: Overall graft survival is defined as not having graft loss (re-transplant, return to dialysis for more than 30 consecutive days, or death) at any time following skin closure. Data is reported as the percentage of patients with Overall Graft Survival.
  End of Study was defined as the last day of evaluation and could have included bivariate assessments after 36 months.
Time Frame: End of Study (36 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 88.6 | 82.6 | 90.9 | 91.2
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.3155, normal approximation; differences in event rates = 6.0, 95% CI 2-sided [-5.7 to 17.6]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p = 0.9045, normal approximation; differences in event rates = -0.4, 95% CI 2-sided [-6.5 to 5.7]

8. Secondary Outcome: Patient Survival at 12 Months
Description: Patient survival is defined as not dead within 12 months after skin closure.
  Kaplan Meier analysis was used to estimate percentage of patients with event. Patients with no event by the time of the scheduled visit or whose first event was after premature discontinuation of randomized study drug or tacrolimus were censored on the scheduled day of assessment, on the day of premature treatment discontinuation or last evaluation day, whichever came first.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 98.6 | 96.9 | 98.1 | 98.7
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.5265, normal approximation; Analysis based on normal approximation using Greenwood's formula for standard error; differences in event rates = 1.6, 95% CI 2-sided [-3.4 to 6.7]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p = 0.6820, normal approximation; Analysis based on normal approximation using Greenwood's formula for standard error; differences in event rates = -0.6, 95% CI 2-sided [-3.4 to 2.2]

9. Secondary Outcome: Overall Patient Survival
Description: Overall patient survival is defined as not dead at any time following skin closure. Data is reported as the percentage of patients with Overall Patient Survival.
  End of Study was defined as the last day of evaluation and could have included bivariate assessments after 36 months.
Time Frame: End of Study (36 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
Percentage of Patients | 95.7 | 89.9 | 93.9 | 95.3
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; Test type: Superiority or Other; p = 0.1797, normal approximation; differences in event rates = 5.9, 95% CI 2-sided [-2.7 to 14.4]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; Test type: Superiority or Other; p = 0.5655, normal approximation; differences in event rates = -1.4, 95% CI 2-sided [-6.3 to 3.4]

10. Secondary Outcome: Renal Function Abnormalities Based on Creatinine Clearance
Description: Increases in creatinine clearance usually indicates an improvement.
  Change in creatinine clearance from month 1 was calculated.
  Change from 1 month is calculated by month 36 - month 1.
Time Frame: 1 month and End of Study (36 months)
Population: The number of participants analyzed represents Full Analysis Set: all patients who were transplanted in the study and received at least 1 dose of tacrolimus and at least 1 dose of study drug. Only patients with the test result at a given time point were included in each time point analysis, and these numbers are noted in the category titles as "N".
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
mL/s
  Month 1 (N= 65; 65; 162; 161) | 0.882 (0.3585) | 0.833 (0.2515) | 0.906 (0.2720) | 0.891 (0.2668)
  Month 36 (N= 48; 47; 125; 131) | 0.976 (0.3772) | 0.862 (0.2929) | 1.011 (0.2736) | 1.039 (0.3195)
  Change from Month 1 (N= 48; 46; 125; 129) | 0.031 (0.3599) | 0.039 (0.2649) | 0.080 (0.2592) | 0.140 (0.2698)
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; P-Value applies to 'Change from Month 1'; Test type: Superiority or Other; p = 0.4735, ANCOVA; Analysis tests the difference between treatment groups for the mean change from month 1 with the month 1 value as covariate
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; P-Value applies to 'Change from Month 1'; Test type: Superiority or Other; p = 0.1186, ANCOVA; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: Renal Function Abnormalities Based on Serum Creatinine
Description: Decrease in serum creatinine usually indicates an improvement.
  Change in creatinine clearance from month 1 was calculated.
  Change from 1 month is calculated by month 36 - month 1.
Time Frame: 1 month and End of Study (36 months)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Number analyzed (Participants) | 70 | 69 | 164 | 171
mcmol/L
  Month 1 (N= 67; 65; 163; 162) | 151.7 (88.12) | 155.9 (97.18) | 139.0 (56.82) | 138.2 (46.03)
  Month 36 (N= 49; 47; 126; 131) | 136.6 (68.38) | 152.0 (84.85) | 121.7 (40.09) | 117.1 (35.50)
  Change from Month 1 (N= 49; 46; 126; 129) | 1.8 (69.41) | 3.4 (92.80) | -8.0 (44.07) | -18.7 (42.35)
Statistical Analysis 1: Comparison: Alemtuzumab High-Risk Patients vs Conventional High-Risk Patients; P-Value applies to 'Change from Month 1'; Test type: Superiority or Other; p = 0.5231, ANCOVA; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Alemtuzumab Low- Risk Patients vs Conventional Low-Risk Patients; P-Value applies to 'Change from Month 1'; Test type: Superiority or Other; p = 0.1220, ANCOVA; [statistical method as in outcome 10, analysis 1]

ADVERSE EVENTS:
Description: Data includes Adverse Events (AEs) that started any time between skin closure and 10 days after the last dose of tacrolimus.
  Within a system organ class patients may have reported more than one type of event.
Arm/Group | Alemtuzumab High-Risk Patients | Conventional High-Risk Patients | Alemtuzumab Low- Risk Patients | Conventional Low-Risk Patients
Serious Adverse Events (participants affected / at risk) | 33/70 | 40/69 | 91/164 | 81/171
Other Adverse Events (participants affected / at risk) | 61/70 | 66/69 | 151/164 | 157/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab High-Risk Patients (N=70) | Conventional High-Risk Patients (N=69) | Alemtuzumab Low- Risk Patients (N=164) | Conventional Low-Risk Patients (N=171)
Pneumonia (Infections and infestations) | 1 | 6 | 6 | 2
Urinary tract infection (Infections and infestations) | 4 | 2 | 4 | 6
Bk virus infection (Infections and infestations) | 2 | 2 | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 3 | 5 | 3
Bacteraemia (Infections and infestations) | 2 | 0 | 2 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 0 | 6 | 2
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1 | 3 | 2
Gastroenteritis (Infections and infestations) | 2 | 0 | 5 | 1
Sepsis (Infections and infestations) | 0 | 2 | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 1 | 1 | 3
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 2
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0 | 2
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 2 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 2 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia aspergillus (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 7 | 3
Viral infection (Infections and infestations) | 0 | 1 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 2 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 0
Orchitis (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 1
Campylobacter intestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Candida osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis gangrenous (Infections and infestations) | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium colitis (Infections and infestations) | 0 | 0 | 1 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Cryptococcosis (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis norwalk virus (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Human polyomavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Pericarditis infective (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonitis cryptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1 | 0
West nile viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 5 | 5 | 7 | 10
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Immunosuppressant drug level increased (Investigations) | 1 | 0 | 0 | 0
Pulmonary function test increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 0
Protein urine present (Investigations) | 0 | 0 | 2 | 0
Bacteria urine identified (Investigations) | 0 | 0 | 1 | 0
Blood culture positive (Investigations) | 0 | 0 | 1 | 0
Cytomegalovirus antigen positive (Investigations) | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 4 | 2 | 6 | 12
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 9
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Renal lymphocele (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Stenosis of vesicourethral anastomosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Treatment noncompliance (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 3 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 6
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 7
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 5
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 2
Aneurysm arteriovenous (Vascular disorders) | 0 | 1 | 0 | 0
Lymphocele (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 3
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 0
Necrosis ischaemic (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 2 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 3 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery atherosclerosis (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 2 | 0 | 2
Death (General disorders) | 0 | 1 | 1 | 0
Heparin-induced thrombocytopenia (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 3
Chills (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 3 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 2 | 0 | 2 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1 | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2 | 6
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 2 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 2 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephritis interstitial (Renal and urinary disorders) | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Parathyroidectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 0 | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 3 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab High-Risk Patients (N=70) | Conventional High-Risk Patients (N=69) | Alemtuzumab Low- Risk Patients (N=164) | Conventional Low-Risk Patients (N=171)
Anaemia (Blood and lymphatic system disorders) | 41 | 41 | 90 | 73
Leukopenia (Blood and lymphatic system disorders) | 38 | 40 | 84 | 48
Neutropenia (Blood and lymphatic system disorders) | 8 | 3 | 23 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 7 | 12 | 4
Diarrhoea (Gastrointestinal disorders) | 23 | 18 | 53 | 65
Nausea (Gastrointestinal disorders) | 8 | 10 | 16 | 11
Vomiting (Gastrointestinal disorders) | 4 | 7 | 12 | 8
BK Viris infection (Infections and infestations) | 3 | 7 | 10 | 9
Bronchitis (Infections and infestations) | 3 | 6 | 8 | 9
Cytomegalovirus infection (Infections and infestations) | 2 | 4 | 11 | 6
Escherichia urinary tract infection (Infections and infestations) | 0 | 2 | 9 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 27 | 23
Urinary tract infection (Infections and infestations) | 18 | 14 | 32 | 37
Urinary tract infection bacterial (Infections and infestations) | 1 | 5 | 5 | 5
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 6 | 12 | 16 | 13
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 4 | 8 | 13
Blood creatinine increased (Investigations) | 7 | 3 | 18 | 14
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 1 | 7 | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 7 | 11 | 11
Hyperlipidaemia (Metabolism and nutrition disorders) | 12 | 16 | 33 | 32
Tremor (Nervous system disorders) | 0 | 1 | 10 | 7
Hypertension (Vascular disorders) | 9 | 7 | 25 | 18

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.